CLINICAL TRIAL: NCT04756401
Title: Open Label, Phase 2, Single-Arm Study of Selinexor, Daratumumab, Carfilzomib and Dexamethasone for High-Risk, Relapsed and Relapsed/Refractory Multiple Myeloma Patients Who Have Received 1 - 3 Prior Lines of Therapy
Brief Title: Selinexor, Daratumumab, Carfilzomib and Dexamethasone for the Treatment of High-Risk, Recurrent or Refractory Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACCRU-MY-1901; NCI-2020-13697 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACCRU-MY-1901 (Other: Academic and Community Cancer Research United); P30CA015083 (NIH)
Record Dates: First submitted 2021-01-04; First posted 2021-02-16 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; daratumumab; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (carfilzomib, daratumumab, dexamethasone, selinexor) (Experimental): Patients receive carfilzomib IV over 30 minutes on days 1, 8, and 15 and daratumumab IV on days 1 and 2 of cycle 1 then days 8, 15, and 22 of cycle 1, then, days 1, 8, 15, and 22 of cycle 2, days 1 and 15 of cycles 3-6, and day 1 of subsequent cycles. Patients also receive dexamethasone PO on days 1, 8 15, and 22, and selinexor PO on days 1, 8, and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carfilzomib; Biological: Daratumumab; Drug: Dexamethasone; Other: Quality-of-Life Assessment; Drug: Selinexor

INTERVENTIONS:
Drug: Carfilzomib — Given IV
  Other Names: Kyprolis; PR-171
Biological: Daratumumab — Given IV
  Other Names: Anti-CD38 Monoclonal Antibody; Darzalex; HuMax-CD38; JNJ-54767414
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Drug: Selinexor — Given PO
  Other Names: ATG-010; CRM1 Nuclear Export Inhibitor KPT-330; KPT-330; Selective Inhibitor of Nuclear Export KPT-330; SINE KPT-330; Xpovio

SUMMARY:
This phase II trial studies the effect of selinexor when combined with carfilzomib, daratumumab, and dexamethasone in treating patients with high-risk multiple myeloma that has come back (recurrent) or has not responded to treatment (refractory) and who have received 1-3 prior lines of therapy. Selinexor may stop the growth of cancer cells by blocking a protein called CRM1 that is needed for cell growth. Carfilzomib is a type of drug called a proteasome inhibitor. A proteasome is a protein found within cells that has the important role of identifying and marking damaged proteins that are needed to be destroyed by the cell for survival. The inhibition of the proteasome allows for damaged protein to accumulate within cells. This accumulation of damaged protein causes the cell to die. Daratumumab is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. Anti-inflammatory drugs, such as dexamethasone lower the body's immune response and are used with other drugs in the treatment of some types of cancer. Giving selinexor in combination with carfilzomib, daratumumab, and dexamethasone may work better than carfilzomib, daratumumab, and dexamethasone alone in treating patients with multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the minimal residual disease (MRD) negativity rate, at 10^-5 level of sensitivity by flow cytometry in bone marrow, with the addition of selinexor to daratumumab, carfilzomib and dexamethasone (SKDd) in patients with high-risk, relapsed or relapsed/refractory multiple myeloma.

SECONDARY OBJECTIVES:

I. To evaluate the overall response rate (partial response [PR] or better) of patients receiving SDKd combination for high risk, relapsed or relapsed/refractory multiple myeloma (MM) and assess depth of response (very good partial response [VGPR], complete response [CR], stringent complete response [sCR]).

II. To evaluate the time to response and duration of response in patients receiving SDKd combination for MM.

III. To evaluate the progression free survival and overall survival in patient receiving SDKd.

IV. To evaluate the MRD negativity rates to the level of sensitivity 10^-6 by flow cytometry in bone marrow.

V. To evaluate the safety profile of the SDKd combination.

CORRELATIVE RESEARCH OBJECTIVES:

I. To explore the impact of baseline immunomodulatory derivative (IMiD)-14 scores gene expression profile (GEP) on progression free survival.

II. Quality of life assessment utilizing Quality of Life Questionnaire (QLQ)-Core (C) 30 and QLQ-Multiple Myeloma (MY) 20 (Cocks et al., 2007; Wisloff et al., 1996).

OUTLINE:

Patients receive carfilzomib intravenously (IV) over 30 minutes on days 1, 8, and 15 and daratumumab IV as a split dose on cycle 1 days 1 and 2 then on days 8, 15, and 22 of cycle 1, then on days 1, 8, 15, and 22 of cycle 2, days 1 and 15 of cycles 3-6, and day 1 of subsequent cycles. Patients also receive dexamethasone orally (PO) on days 1, 8 15, and 22, and selinexor PO on days 1, 8, and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients without disease progression/clinical relapse or have initiated subsequent anti-cancer therapy, are followed up every 3 months until progression/clinical relapse or initiation of subsequent anti-cancer therapy, and then every 6 months for up to 5 years. Patients with disease progression/clinical relapse or have initiated subsequent anti-cancer therapy are followed up every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Patients must have a documented history of relapsed or relapsed/refractory MM as defined by International Myeloma Working Group (IMWG) criteria (Rajkumar et al., 2014)

  * Patients must be selinexor and carfilzomib sensitive
  * Prior daratumumab exposure is allowed, provided that it has been 6 months or more from the time of cycle 1 day 1 (C1D1) of protocol therapy
* High risk disease defined as 1 or more of the following:

  * High risk cytogenetics (any of the following)

    * t(4;14), t(14;16), t(14;20)
    * del(17p)
    * del(1p)
    * Gain 1q (>= 3 copies)
  * Lactate dehydrogenase (LDH) > upper limit of normal at relapse
  * International Staging System (ISS) stage 3 disease at relapse
  * Extramedullary disease at diagnosis or relapse
  * >= 5% circulating plasma cells at diagnosis or relapse
  * High risk by gene expression profiling, if known, at diagnosis or relapse
  * Early relapse with first-line therapy

    * =< 18 months from cycle 1 day 1 for patients not undergoing autologous stem cell transplant (ASCT)
    * =< 36 months from cycle 1 day 1 for patients undergoing ASCT and post-ASCT maintenance
* Measurable disease
* 1-3 prior lines of therapy
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) =< 2 (Form is available on the Academic and Community Cancer Research United [ACCRU] website)
* Patients must have evidence of adequate bone marrow reserves, as defined by the following:

  * Absolute neutrophil count (ANC) >= 1,000 cells/mm^3 without filgrastim or its equivalent within 1 week of the initiation of treatment or pegfilgrastim or its equivalent within 2 weeks of the initiation of treatment
  * Platelet count of >= 100,000 cells/mm^3 for patients who have bone marrow plasmacytosis of < 50%, or >= 50,000 cells/mm^3 for patients who have bone marrow plasmacytosis of > 50%, both without platelet transfusion support within 1 week of the initiation of treatment or the use of TPO mimetics
  * NOTE: If your site laboratory reports use different units of measurements than what is required by the protocol eligibility requirements, please use the "Lab Test Unit Conversion Worksheet" available on the ACCRU website under "General Forms"
* Total bilirubin =< 2.0 times the upper limit of the institutional normal values except in subjects with congenital bilirubinemia, such as Gilbert syndrome (in which case a direct bilirubin =< 1.5 x upper limit of normal [ULN] is required)
* Total aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 times the upper limit of the institutional normal values
* Patients must have adequate cardiac function defined as left ventricular ejection fraction (LVEF) >= 45% by echocardiogram, magnetic resonance imaging (MRI) or multigated acquisition (MUGA) scan
* For those with symptomatic pulmonary disease (e.g. chronic obstructive pulmonary disease [COPD], asthma) or other signs/symptoms of pulmonary disease, adequate pulmonary function as defined by a forced expiratory volume in one second (FEV1) >= 50% of predicted and diffusing capacity for carbon monoxide (DLCO)/alveolar volume (VA) >= 50% of predicted within 28 days prior to day 1 of treatment

  * Note: Baseline pulmonary function tests are only required on an as needed basis
* Patients must have evidence of adequate renal function, as defined by the following: creatinine clearance (CrCl) >= 30 mL/min., as measured by a 24-hour urine collection, or estimated by the Cockcroft and Gault formula

  * Calculated creatinine clearance must be >= 30 ml/min using the Cockcroft-Gault formula
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Female patients of childbearing potential must have a negative serum pregnancy test at screening and agree to use highly effective (dual methods of) contraception throughout the study and for 6 months following the last dose of study drug; and male patients must use an effective barrier method of contraception throughout the study and for 3 months following the last dose of study drug if sexually active
* Ability to complete questionnaire(s) by themselves or with assistance
* Provide informed written consent =< 28 days prior to registration
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)

Exclusion Criteria:

* Prior treatment with daratumumab within 6 months from cycle 1 day1
* Patient with carfilzomib-refractory disease defined as disease progression on or within 60 days of last carfilzomib dose
* Any of the following because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Uncontrolled hypertension, defined as a systolic blood pressure of >= 160 mmHg or a diastolic blood pressure of >= 90 mmHg
* Significant cardiac disease, including any of the following:

  * >= class 3 New York Heart Association (NYHA) congestive heart failure
  * Electrocardiogram (EKG) evidence of acute ischemia
  * Unstable angina
  * Myocardial infarction within 6 months prior to day 1 of treatment
  * Clinically significant arrhythmias or conduction block (premature atrial contractions [PACs], premature ventricular contractions [PVCs], rate controlled atrial fibrillation, sinus arrhythmia, asymptomatic sinus bradycardia or sinus tachycardia and 1st degree heart block are not considered clinically significant)
  * >= grade 2 QT interval by Fridericia (QTcF) prolongation (i.e. > 480 ms)
  * Note: Prior to study entry, any EKG abnormality at screening not felt to put the patient at risk must be documented by the investigator as not medically significant
* A diagnosis of human immunodeficiency virus (HIV) does not exclude the patient from participation. However, the viral load must be < 50 copies/mm^3 and CD4 count >= 200 on anti-HIV therapy within 28 days prior to cycle 1, day 1 of treatment
* Positive hepatitis C antibody test result or positive hepatitis C ribonucleic acid (RNA) test result at screening

  * NOTE: Subjects with positive hepatitis C antibody due to prior eradicated disease can be enrolled if a confirmatory negative hepatitis C RNA test is obtained
* Is seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Subjects with resolved infection (i.e. subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) deoxyribonucleic acid (DNA) levels. Subjects who are PCR positive will be excluded. Exception: patients with serologic findings suggestive of HBV vaccination
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements
* Discontinuation of prior carfilzomib or daratumumab due to treatment toxicity
* Radiation within 14 days prior to day 1 of treatment. Note: palliative radiation therapy (XRT) to < 5% of the total marrow volume as assessed by the treating investigator is allowed within 14 days
* Major surgery within 4 weeks prior to day 1 of treatment
* Any multiple myeloma therapy within 14 days prior to cycle 1, day 1
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Active central nervous system (CNS) involvement
* Concomitant amyloid light-chain (AL) amyloidosis or polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes (POEMS) syndrome
* Patients cannot have other prior or concomitant malignancies except for:

  * Non-melanoma skin cancer
  * In situ malignancy
  * Low-risk prostate cancer after curative therapy
  * Prostate cancer Gleason grade 6 AND with stable prostate specific antigen (PSA) levels off treatment
  * Other cancer for which the patient has been treated with curative intent or disease free for >= 3 years
* Prior exposure to daratumumab within 24 weeks from cycle 1, day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-12-08 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of minimal residual disease (MRD) negative status | Up to 5 years post-treatment
  MRD negative status at 10^-5 level of sensitivity by flow cytometry will be considered synonymous with "success", unless specified otherwise. The proportion of success will be estimated by the number of success divided by the total number of evaluable patients. 95% confidence intervals for the true success proportion will be calculated according to the approach of Duffy and Santner.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 5 years post-treatment
  Will be estimated by the total number of patients who achieve a confirmed response at any time divided by the total number of evaluable patients. A confirmed response is defined as a partial response (PR), very good partial response (VGPR), complete response (CR) or stringent complete response (sCR) noted as the objective status on two consecutive evaluations at least two weeks apart. Exact binomial 95% confidence intervals for the true overall response rate will be calculated. The depth of response (PR versus VGPR versus CR versus sCR) will also be summarized.
Time to response | Time between registration and earliest date of documentation of response using International Myeloma Working Group criteria, assessed up to 5 years
  Time to response (TTR) is defined as time from the date of registration to the date of confirmed response using IMWG criteria. TTR will be summarized descriptively (median, range).
Duration of response | Time between first documentation of response to the earliest date of progression or death, assessed up to 5 years
  Duration of response (DOR) is defined as time from date at which the patient's confirmed objective status is noted to the earliest date of progression or death. The DOR will be estimated using the method of Kaplan-Meier.
Progression-free survival | Time between registration to the earliest date of documentation of disease progression or death due to any cause, assessed up to 5 years
  The progression free survival (PFS) is defined as the time from registration to the earliest date of documentation of disease progression or death due to any cause. The distribution of PFS will be estimated using method of Kaplan-Meier.
Overall survival (OS) | Time between registration to death due to any cause, assessed up to 5 years
  The overall survival (OS) is defined as the time from registration to death due to any cause. The distribution of OS will be estimated using method of Kaplan-Meier.
MRD negativity rate at 10^-6 of sensitivity | Up to 5 years post-treatment
  Will be assessed in the bone marrow by flow cytometry estimated as the number of patients who have achieved MRD negative result at 10^-6 level of sensitivity at any time divided by the total number of evaluable patients. Exact 95% binomial confidence intervals for the true rate of MRD negative response will also be calculated.
Incidence of adverse events | Up to 30 days after the last dose of study drug or until the start of subsequent antineoplastic therapy, whichever occurs first
  Will be assessed per National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the adverse events to the study treatment will be taken into consideration.

OTHER OUTCOMES:
Effect of Immunomodulatory imide drug-14 scores gene expression profile (GEP) on Progression-Free Survival | Baseline up to progression-free survival, assessed up to 5 years
  The progression free survival (PFS) is defined as the time from registration to the earliest date of documentation of disease progression or death due to any cause. Patients will be categorized by their GEP and progression-free survival estimates will be compared across GEP scores.
Change in EORTC QLQ-C30 scores from baseline to end of treatment | Baseline up to progression, withdrawal, or end of treatment, assessed up to 5 years
  QOL will be measured using the EORTC QLQ-C30, a patient-reported questionnaire about patient ability to function, symptoms related to the cancer and its treatment, overall health and quality of life, and perceived financial impact of the cancer and its treatment. Changes in raw score from baseline to end of treatment will be assessed, in each of the physical and mental health domains. The Wilcoxon signed-rank test will be utilized to assess changes in raw scores. Mean change, along with standard deviation will be reported.
Change in EORTC QLQ-MY20 scores from baseline to end of treatment | Baseline up to progression, withdrawal, or end of treatment, assessed up to 5 years
  QOL will be measured using the QLQ-MY20, a patient-reported questionnaire about patient ability to function, symptoms related to the cancer and its treatment, overall health and quality of life, and perceived financial impact of the cancer and its treatment. Changes in raw score from baseline to end of treatment will be assessed, in each of the physical and mental health domains. The Wilcoxon signed-rank test will be utilized to assess changes in raw scores. Mean change, along with standard deviation will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Shebli Atrash, Principal Investigator — Academic and Community Cancer Research United
Locations (4):
- United States (4):
  - Hackensack University Medical Center, Hackensack, New Jersey
  - State University of New York Upstate Medical University, Syracuse, New York
  - UNC Lineberger Comprehensive Cancer Center University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina